CLINICAL TRIAL: NCT04171934
Title: Clinical Validation of a Video-based Epilepsy Examination Service
Acronym: Nelli
Status: Completed | Type: Observational
Sponsor: Tampere University (Other)
Collaborators: Filadelfia Epilepsy Hospital (Other); Aarhus University Hospital (Other); Neuro Event Labs Oy (Unknown)
Responsible Party: Principal Investigator, Jukka Peltola, Professor, Department of Neurology, Tampere University
Other Study IDs: CS001
Record Dates: First submitted 2019-11-12; First posted 2019-11-21 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Epilepsy; Seizure
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults: Subjects 22+ years of age
- Pediatric: Subjects less than 22 years of age

SUMMARY:
The main purpose of this study is to validate the ability of the Nelli system (video-based epilepsy examination system) to detect epileptic motor seizure behaviors in patients at rest.

DETAILED DESCRIPTION:
Proper seizure documentation is an important tool to evaluate treatment outcomes and risks associated with epileptic seizures. Apart from a costly in-hospital video electro-encephalogram (VEEG) monitoring, most patients with epilepsy log and track their seizures with the help of the seizure diaries only. However, the reliability of the diaries is heavily dependent on an accurate recognition and recording of the seizures. There is an obvious need for a more objective and reliable seizure detection method. The investigators propose a low-cost video-based examination system, designed to detect motor seizure behaviors in patients at rest.

The main aim of this study is to clinically validate the ability of the Nelli system (video-based epilepsy examination system) to detect epileptic motor seizure behaviors in patients at rest, using simultaneous VEEG as the ground truth with the reference to all motor seizures and individual motor seizure types.

Study design established as follows:

1. Study population is represented by 90 epilepsy patients with suspected history of motor seizures undergoing a standard VEEG examination for clinical evaluation of epilepsy.
2. Co-registration of standard VEEG with the Nelli video- and audio-based system is performed, duration of the registration is 1-4 days.
3. The inclusion criteria for seizures:

   1. Epileptic motor seizures appearing from rest while patients are in supine position in their monitoring bed.
   2. The seizures are determined to be epileptic based on electroclinical characteristics by the responsible neurophysiologist / epileptologist.
   3. The seizures can be classified into motor seizure types (both focal and generalized) using the 2017 International League Against Epilepsy (ILAE) seizure classification.
4. The registrations are analyzed by the Nelli system blinded to any clinical information. Nelli system consists of two evaluation components:

   1. Algorithmic component (pre-trained machine learning model based on video and audio signals)
   2. Supervisory component (performed by experienced VEEG technicians)
5. Reports containing the seizure type classification (time-stamped) are provided by the VEEG laboratory, the performance of the Nelli system is assessed using these reports as the ground truth.

   a. Specificity and sensitivity of the Nelli system are evaluated with reference to both all motor seizures and individual motor seizure types.
6. The secondary outcome measures are established as follows:

   1. To assess the latency from the onset of the seizure detection by the Nelli system in comparison to VEEG registration.
   2. To determine an inter-rater agreement for the supervisory component of the Nelli system.
   3. To investigate the performance of the algorithmic component of the Nelli system alone.

ELIGIBILITY:
Inclusion Criteria:

Patients with epilepsy undergoing a standard VEEG examination for clinical evaluation consenting to participate in the present study

Exclusion Criteria:

Patients not consenting to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 90 epilepsy patients of various ages undergoing a standard VEEG examination for clinical evaluation in either one of the following medical facilities: Danish Epilepsy Center (Filadelfia) or Aarhus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
FDR (per hour) and TPR | Examination period specific to the patient (1-4 days)
  False detection rate (FDR/hour) as well as true positive rate (TPR) of the Nelli service is to be evaluated. Here FDR stands for detections which do not intersect with the ground truth events, and true positive events match ground truth with the Nelli detections.

SECONDARY OUTCOMES:
Latency (seconds) | Examination period specific to the patient (1-4 days)
  Latency from the seizure onset (according to the ground truth) and the seizure detection by the Nelli system.
Inter-rater agreement (Cohen's kappa coefficient) | Examination period specific to the patient (1-4 days)
  Inter-rater agreement for the supervisory component of the Nelli system
Performance of the algorithmic component | Examination period specific to the patient (1-4 days)
  Performance of the algorithmic component evaluated using the ROC (receiver operating characteristic) curve at different operating points (thresholds).

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Epilepsy Center, Filadelfia, Dianalund, Denmark